CLINICAL TRIAL: NCT03304132
Title: The Oral Microbiome and Upper Aerodigestive Squamous Cell Cancer
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-01834
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Oral Cancer
Keywords: Oral Microbiome; reflux disorders; esophageal microbiome; Alcohol Use; Tobacco Use
MeSH Terms: conditions — Mouth Neoplasms; Alcohol Drinking; Tobacco Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 140 UADSCC cases and 420 controls using Roche 454 16S rRNA gene sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Upper aerodigestive squamous cell cancers (UADSCC) cases: From PLCO and ACS CPS II, identified 140 UADSCC cases. These cases are frequency matched 3:1 (420 controls) by incidence density sampling for study (ACS. PLCO),
  Interventions: Other: Classification of Oral Microbiome Using 16S rRNA gene sequence-based approach; Other: Classification of Oral Microbiome Using taxonomic approach
- Controls: From PLCO and ACS CPS II, we have identified 140 UADSCC cases. These cases are frequency matched 3:1 (420 controls) by incidence density sampling for study (ACS. PLCO),
  Interventions: Other: Classification of Oral Microbiome Using 16S rRNA gene sequence-based approach; Other: Classification of Oral Microbiome Using taxonomic approach

INTERVENTIONS:
Other: Classification of Oral Microbiome Using 16S rRNA gene sequence-based approach — The sequence-based approach is selected because it classifies samples by considering the entire difference (genetic distance) in 16S rRNA gene sequences among samples analyzed, unbiased by artificial details such as taxonomies, sequence length, or even quality scores.
Other: Classification of Oral Microbiome Using taxonomic approach — The taxonomic approach is a complement to the sequence-based approach in that it will further identify specific taxonomic groups or species that can explain the difference found by overall analyses.

SUMMARY:
The human oral cavity is a diverse habitat that contains approximately 700 prokaryotic species. The oral microbiome is comprised of 44% named species, 12% isolates representing unnamed species, and 44% phylotypes known only from 16S rRNA based cloning studies (http://www.homd.org/). Species from 11 phyla have been identified: Firmicutes, Bacteroidetes, Proteobacteria, Actinobacteria, Spirochaetes, Fusobacteria, TM7, Synergistetes, Chlamydiae, Chloroflexi and SR1 (http://www.homd.org/). Because these observations have been mainly based on data generated from traditional Sanger sequencing, the diversity of oral microbiome is highly likely underestimated. Application of high throughput sequencing to the oral microbiome similar to the scale of the microbiome studies of other body sites (GI tract, skin, and vagina) under the Human Microbiome Project is necessary to obtain data essential for understanding the diversity and community structure of the oral microbiome in health and disease.

DETAILED DESCRIPTION:
The Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Trial and The American Cancer Society Cancer Prevention Study II (CPS-II) investigators have identified 140 UADSCC cases that have been frequency matched 3:1 (420 controls) by incidence density sampling for study (ACS. PLCO), gender, ethnic background, and age, within 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Upper Aerodigestive Squamous Cell Cancer and registered in:
* The American Cancer Society Cancer Prevention Study II (CPS-II)
* The Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Trial.

Ages: 40 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The American Cancer Society Cancer (ACS) Prevention Study II Nutrition Cohort (CPS-II) was established in 1992; the cohort includes over 86,000 men and 97,000 women from 21 U.S. states who completed a mailed questionnaire in 1992. In total, 72 UADSCC were eligible for study, with completed informed consent and prediagnostic oral wash collection.
  The Prostate, Lung, Colon and Ovarian (PLCO) Cancer Screening Trial is a randomized controlled trial of approximately 155,000 men and women. Participants are randomized to either a screening or control arm. n total, 68 UADSCC were eligible for study, including completed informed consent and prediagnostic oral wash collection.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 1992-12-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
16S rRNA gene survey approach for microbiome characterization | 4 Years
  Data alignment and clustering to determine microbiome species diversity

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Ahn, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No